CLINICAL TRIAL: NCT03366961
Title: The Multi-national Multi-institutional Phase 2 Trial for Conversion Surgery in Stage IV or Unresectable Gastric Cancer
Brief Title: Conversion Surgery in Stage IV or Unresectable Gastric Cancer
Acronym: ConGC-II
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Cho Hyun Park (Other)
Collaborators: The Catholic University of Korea (Other); Peking University (Other)
Responsible Party: Sponsor-Investigator, Cho Hyun Park, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ConGC-II
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Stage IV or Unresectable Gastric Cancer
MeSH Terms: interventions — Conversion to Open Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conversion surgery (Other): Palliative chemotherapy followed by radical gastrectomy
  Interventions: Procedure: Conversion surgery

INTERVENTIONS:
Procedure: Conversion surgery — Palliative chemotherapy followed by radical gastrectomy

SUMMARY:
This study aims to identify the safety and the survival benefit of the conversion surgery in stage IV or unresectable gastric cancer. The study designed single-arm phase II trial. All the patients would undergo curative-intent radical gastrectomy after palliative chemotherapy if the tumor responded to the chemotherapy. Primary endpoint was three-year overall survival. Secondary endpoints included short-term postoperative outcomes within 30 days, three-year relapse free survival, and success rate of conversion surgery (rate of R0 resection).

DETAILED DESCRIPTION:
The survival rate of patients with stage IV gastric cancer (GC) is very low. Recently, several retrospective studies about conversion surgery have been introduced. The results of the studies showed around 30~40% of three-year survival rate in conversion surgery group. Eight institutions in Catholic University of Korea analyzed 419 stage IV GC patients, and they had divided into four groups: chemotherapy only, chemotherapy followed by gastrectomy, gastrectomy followed by chemotherapy, and best supportive care group. The group of gastrectomy followed by chemotherapy, which is similar with conversion surgery, showed 40% of three-year survival rate. However, the study included only small number of patients who were in conversion surgery group, and had several biases. Thus, we planned multi-national, multi-center phase II trial for conversion surgery in stage IV or unresectable GC.

ELIGIBILITY:
Inclusion Criteria:

* Gastric adenocarcinoma
* Stage IV or unresectable gastric cancer was diagnosed by pre-operative evaluation including endoscopy, endoscopic ultrasound, Computed tomography (CT), Positron emission tomography-computed tomography (PET CT), or staging laparoscopy
* Partial or complete response to chemotherapy
* Eastern Cooperative Oncology Group (ECOG) score <3
* Who agreed to enroll the study

Exclusion Criteria:

* Synchronous or metachronous malignancy
* remnant gastric cancer
* BMI less than 18.5
* Pregnancy

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival | 3 years after the surgery
  3-year overall survival after conversion surgery

SECONDARY OUTCOMES:
Complication | 30 days after the surgery
  Short-term complication rate after conversion surgery
3-year disease free survival | 3 years after the surgery
  3-year disease free survival after conversion surgery
Success rate of conversion surgery | 30 days after the surgery
  Rate of R0 resection
Response rate of chemotherapy | Operation day
  Response rate of chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea